CLINICAL TRIAL: NCT06883825
Title: Temporomandibular Joint Respiratory and Thoracic Region Added to Myofunctional Rehabilitation in Dysfunction Comparison of the Effects of Exercises: A Randomized Controlled Trial
Brief Title: Temporomandibular Joint Respiratory and Thoracic Region Added to Myofunctional Rehabilitation in Dysfunction Comparison of the Effects of Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merve Keskin (Other)
Responsible Party: Sponsor-Investigator, Merve Keskin, Research Assisstant, Izmir Katip Celebi University
Organization: Izmir Katip Celebi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0090
Record Dates: First submitted 2025-02-24; First posted 2025-03-19 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-02

CONDITIONS: Temporomandibular Joint Dysfunction; Myofunctional Therapy; Rehabilitation Exercise
Keywords: temporomandibular joint dysfunction; myofunctional therapy; rehabilitation; exercise; thoracic region; diapragmatic breathing
MeSH Terms: conditions — Temporomandibular Joint Disorders; Motor Activity | interventions — Myofunctional Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Myofunctional Therapy (Active Comparator): Participants will only receive myofunctional rehabilitation therapy. This treatment includes massage and exercises to improve the function of the jaw muscles.
  Interventions: Other: Myofunctional Therapy
- Myofunctional Therapy + Respiratory Exercises (Experimental): Participants will receive breathing exercises as well as myofunctional therapy. This treatment includes exercises to improve jaw function and support the respiratory system.
  Interventions: Other: Myofunctional Therapy + Respiratory Exercises
- Myofunctional Therapy + Thoracic Region Exercises (Experimental): Participants will receive myofunctional therapy as well as exercises for the thoracic region. This treatment includes exercises to improve jaw function and increase the flexibility of the chest area.
  Interventions: Other: Myofunctional Therapy + Thoracic Region Exercises

INTERVENTIONS:
Other: Myofunctional Therapy — Participants will only receive myofunctional rehabilitation therapy. This treatment includes massage and exercises to improve the function of the jaw muscles.
  Arms: Myofunctional Therapy
Other: Myofunctional Therapy + Respiratory Exercises — Participants will receive breathing exercises as well as myofunctional therapy. This treatment includes exercises to improve jaw function and support the respiratory system.
  Arms: Myofunctional Therapy + Respiratory Exercises
Other: Myofunctional Therapy + Thoracic Region Exercises — Participants will receive myofunctional therapy as well as exercises for the thoracic region. This treatment includes exercises to improve jaw function and increase the flexibility of the chest area.
  Arms: Myofunctional Therapy + Thoracic Region Exercises

SUMMARY:
In the study, a questionnaire form will be applied to the participants using a face-to-face interview technique. Through the questionnaires, demographic characteristics, pain intensity, location of pain, symptoms of dysfunction, oral habits, and loss of function in the jaw joint will be evaluated. Soft tissue (muscle) affections, spine structure, and mobility will be evaluated and recorded in the questionnaire form to be used for the evaluation of jaw joint dysfunctions. Pain level, depression, stress, anxiety level, and sleep quality will be evaluated with the help of a questionnaire.

The aims of this study were;

1. To investigate the effects of muscle and function therapy on dysfunction, spinal structure and mobility, depression, stress, anxiety, and sleep quality in patients with jaw joint dysfunction,
2. To investigate the effects of breathing exercises added to muscle and function therapy on dysfunction, spine structure and mobility, depression, stress, anxiety, and sleep quality in patients with jaw joint dysfunction,
3. To investigate the effects of back exercises added to muscle and function therapy on dysfunction, spinal structure and mobility, depression, stress, anxiety and sleep quality in patients with jaw joint dysfunction,
4. To compare the effects of muscular and functional therapy alone, respiratory exercises added to muscular and functional therapy, and back exercises on dysfunction, spinal structure and mobility, depression, stress, anxiety, and sleep quality in patients with jaw joint dysfunction.

Hypotheses of this study; H1: Myofunctional rehabilitation in patients with temporomandibular joint dysfunction positively affects TMD dysfunction findings, spinal structure and mobility, and psychosocial effects.

H2: Respiratory exercises added to myofunctional rehabilitation in patients with temporomandibular joint dysfunction have a positive effect on TMD dysfunction findings, spinal structure and mobility, and psychosocial effects.

H3: Thoracic exercises added to myofunctional rehabilitation in patients with temporomandibular joint dysfunction have a positive effect on TMD dysfunction findings, spinal structure, mobility, and psychosocial effects.

H4: In patients with temporomandibular joint dysfunction, only myofunctional rehabilitation, respiratory exercises added to myofunctional rehabilitation, and thoracic exercises have no superiority over each other on TMD dysfunction symptoms, spinal structure mobility, and psychosocial effects.

In the study, a questionnaire form will be applied to the participants usinga face-to-face interview. Through the questionnaires, demographic characteristics, pain intensity, pain location, symptoms of dysfunction, oral habits, and the presence of jaw joint dysfunctions will be evaluated. Soft tissue (muscle) affections, spine structure, and mobility will be assessed and recorded in the questionnaire form to be used for the evaluation of jaw joint dysfunctions. Pain level, depression, stress, anxiety level, and sleep quality will be evaluated with the help of a questionnaire. The evaluation will take approximately 40-45 minutes.

Group 1 will be given a massage to relax the masticatory muscles and exercises for the masticatory muscles and the muscles in the neck region.

The 2nd group will be given breathing exercises in addition to the 1st group. The 3rd group will be given back exercises in addition to the 1st group. One session will last approximately 45-50 minutes, and a total of 16 sessions of treatment will be applied in 8 weeks, 2 sessions per week. Measurements will be taken twice, at the beginning and the end of the 8th week.

DETAILED DESCRIPTION:
This research is planned as a randomized controlled study. The study will be conducted at Izmir Kâtip Çelebi University within two years after ethics committee permission is obtained. The population of the study consists of patients with temporomandibular joint dysfunction. The sample of our study will consist of patients aged 18-65 years with muscle and joint involvement according to the Temporomandibular Disorders Research Diagnostic Criteria, who volunteered to participate in the study. No suitable article using similar methods for calculating the sample size of the study was found. According to the power analysis for two-way analysis of variance in repeated measures using G*Power Version 3.1.9.2 (Franz Faul, Universitat Kiel, Germany) program, the effect size was calculated as f=0.5, number of repetitions=2, number of groups=3, correlation between repeated measures =0.5, Type I error=0.05 and statistical power=0.95, with at least 17 in each group and a total of 51 patients as the number of units in the sample. Considering possible data losses, the number of participants was added by 20% and it was planned to include at least 21 patients in a group and 63 patients in total.

Participants will be divided into three groups as myofunctional rehabilitation group, respiratory exercise group, and thoracic exercise group by block randomization method. Block randomization will be done via https://www.sealedenvelope.com/simple-randomiser/v1/lists.

1st group; deep friction massage to trigger points in masseter and temporalis muscles, mobilization to TMJ and surrounding soft tissues, Rocabodo exercises (6x6), suboccipital relaxation, stretching exercises to upper trapezius, pectoralis minor, levator scapula muscles will be applied.

Group 2 will be given progressive diaphragmatic breathing exercises in addition to group 1. Progression in diaphragmatic breathing exercises will be achieved by adapting the phases of sensorimotor training (static, dynamic, functional) adapted to exercise programs in order to prevent injuries and to ensure strength and stability (15,16).

Diaphragmatic exercises

1. Static Phase (weeks 1-2): It is aimed to provide short-speed motor control and to create kinesthetic awareness. It will include exercises to provide diaphragmatic breathing at each stage of neurodevelopmental steps (supine, side lying, quadripedal, bipedal).
2. Dynamic Phase (weeks 3-5): Following the teaching of diaphragmatic breathing at each stage of neurodevelopmental steps, limb movements will be included in the program with elastic resistance training. In order to teach conscious motor control of movement, they will be asked to maintain diaphragmatic breathing while performing coordinated limb movements at high speeds in a multi-planar field.

3rd Functional Phase (weeks 6-8): After the combination of diaphragmatic breathing with limb movements, exercises including functional complex training on unstable floors will take place in this phase in order to teach the subconscious control of the movement with the progressive resistances of elastic resistance training. For this purpose, elastic resistance bands and exercise balls will be used.

Diaphragmatic breathing exercises will consist of 3 sets of 10 repetitions in each session.

The 3rd group will be given progressive thoracic exercises in addition to the 1st group. Thoracic exercises will consist of 6 exercises including thoracic stretching and mobility exercises lasting 15-20 minutes. Progression in the program will be achieved by changing the color of the elastic resistance band used during the exercises and gradually increasing the number of repetitions of the exercises. To determine the resistance of the elastic resistance band, the participant will be asked to perform the determined movement for 15 repetitions. If the participant's fatigue is at the level of 12-14 (moderate difficulty) according to the Borg scale, which is a subjective questioning tool, it will indicate the appropriate color. Elastic resistance bands are ordered from easy level to more difficult level with skin, yellow, red, green, blue, black, gray, and golden yellow colors.

Exercises for the thoracic region;

1. Thoracic spine extension exercise with a foam roller (2x10),
2. Thoracic extension flexibility exercise (2x10),
3. Thoracic spine rotation exercise (2x8),
4. Thoracic rotation exercise in quadripedal position (2x8),
5. Thoracic rotation exercise in side lying (Open book 2x8),
6. Bird-dog exercise (2x8). One session will last approximately 45-50 minutes, 2 sessions per week, for a total of 16 sessions in 8 weeks. Measurements will be taken twice, at the beginning and the end of the 8th week.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old,
* According to the Temporomandibular Disorders Research Diagnostic Criteria;

  * With muscle involvement,
  * With muscle+joint involvement
* Those who volunteer to participate in the study will be included

Exclusion Criteria:

* According to the Temporomandibular Disorders Research Diagnostic Criteria;
* Those with disc displacement without reduction,
* Those with arthritis
* Those with a known neurological, systemic or psychological disease,
* Pregnant and lactating women,
* Those who have had any trauma/surgical operation in the last 6 months,
* Those with severe to severe local and/or general musculoskeletal pain,
* Patients with an obstructive or restrictive respiratory problem,
* Those with scoliosis that may cause respiratory problems will not be included

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of Temporomandibular Joint Dysfunction | At baseline and from enrollment to the end of treatment at week 8
  Diagnosis of TMD - Evaluated using the Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD), reported as categorical data (diagnosis classification).
Pain Assessment | At baseline and from enrollment to the end of treatment at week 8
  Measured using the Visual Analog Scale (VAS), reported in centimeters (cm)
Symptom Severity | At baseline and from enrollment to the end of treatment at week 8
  Assessed with the Symptom Questionnaire for Temporomandibular Disorders, reported in units on a scale.
Oral Habits Frequency | At baseline and from enrollment to the end of treatment at week 8
  Measured with the Oral Habits Checklist, reported in units on a scale.
Jaw Function Limitation | At baseline and from enrollment to the end of treatment at week 8
  Assessed using the Jaw Function Restriction Scale, reported in units on a scale.
Soft Tissue Examination | At baseline and from enrollment to the end of treatment at week 8
  Assessed using ultrasound to measure masseter muscle thickness and elastography at rest and during contraction, reported in millimeters (mm) and kilopascals (kPa), respectively.

SECONDARY OUTCOMES:
Head Position | At baseline and from enrollment to the end of treatment at week 8
  Measured as the angle between the head and neck, recorded in degrees (°).
Thoracic Region Evaluation | At baseline and from enrollment to the end of treatment at week 8
  Assessed using the Valedo Shape device, with angular measurements recorded in degrees (°).
Thoracic Rotation | At baseline and from enrollment to the end of treatment at week 8
  Measured using a mobile application, recorded in degrees (°).
Depression, Anxiety, and Stress | At baseline and from enrollment to the end of treatment at week 8
  Assessed using the DASS-21 questionnaire, reported in units on a scale.
Sleep Quality | At baseline and from enrollment to the end of treatment at week 8
  Evaluated using a single-item sleep quality scale, reported in units on a scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Celebi University, Çiğli, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No